CLINICAL TRIAL: NCT03925532
Title: A Phase II Multicenter, Single Arm, Open-Label Trial to Evaluate the Efficacy and Safety of Denosumab in Treatment of Post-Allogenic Hematopoietic Stem Cell Transplant Bone Loss
Brief Title: Denosumab in Treating Patients With Bone Loss Due to Donor Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I 78618; NCI-2019-01921 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 78618 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2019-04-16; First posted 2019-04-24 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation Recipient; Osteopenia; Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Supportive Care (denosumab) (Experimental): Patients receive 2 doses of denosumab SC between days 70-130 and days 250-310 after allogeneic hematopoietic stem cell transplant in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Denosumab

INTERVENTIONS:
Biological: Denosumab — Given SC
  Other Names: AMG 162; AMG-162; Prolia; Xgeva

SUMMARY:
This Phase II trial studies the side effects of denosumab and to see how well it works in treating patients with bone loss who have received a donor stem cell transplant. Patients receiving a donor stem cell transplant may experience accelerated bone loss and an increase risk of bone fractures, leading to a decrease in satisfaction and quality of life. A type of immunotherapy drug called denosumab binds to a protein called RANKL, which may help keep bone from breaking down.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy and safety of denosumab therapy for the treatment of bone loss in patients who have received an allogeneic hematopoietic stem cell transplant.

OUTLINE:

Patients receive 2 doses of denosumab subcutaneously (SC) between days 70-130 and days 250-310 after allogeneic hematopoietic stem cell transplant in the absence of disease progression or unacceptable toxicity.

After completion of study treatment patients are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* The patient has undergone an Allogeneic Hematopoietic Stem Cell Transplant
* The patient has completed a base line dual x-ray absorptiometry (DXA) scan =< 6 months prior to transplantation
* The patient has completed a post-transplant DXA scan at day 100 (+/- 30 days) or up to 6 months post transplantation
* The patient has completed and passed a dental clearance exam up to 6 months prior to transplant or 6 months after transplant
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* The patient has a history of a hypersensitivity reaction to denosumab
* The patient has a history of osteonecrosis of the jaw
* The patient has predisposing risk factors for hypocalcemia including the following:

  * Hypoparathyroidism
  * Creatinine clearance (CrCl) < 30 mL/min
  * Dialysis
  * Malabsorption syndrome
* The patient has history of any bone fracture =< 30 days prior to denosumab therapy
* Pregnant or nursing female patients.
* The patient has clinically significant GVHD leading to hospitalization at the time of denosumab dose per prescriber discretion.
* The patient has clinically significant infection leading to hospitalization at the time of denosumab dose (excluding hospitalization due to complexity of treatment leading to inability to treat outpatient, ie. Foscarnet) per prescriber discretion
* The patient is unwilling or unable to follow protocol requirements
* The patient has any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug including relapsed malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip L McCarthy, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Cleveland Clinic, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supportive Care (Denosumab)
Started | 30
Completed | 29
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Supportive Care (Denosumab)
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.38 (9.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Total Hip Percent Change in Bone Mineral Density (BMD)
Description: Day 0 dual x-ray absorptiometry (DXA) scan and day 465 DXA scan will be compared based on the percent change in BMD in the Total hip in allogeneic HSCT patients who have experienced either at least 5% BMD loss between baseline (pre- HSCT) and day + 100 post-HSCT, or who have osteopenia or osteoporosis at either the pre-bone marrow transplant or day + 100 DXA scan.
Time Frame: At baseline and 465 days post-HSCT
Population: All treated and eligible patients that had measures at day 0 and day 465
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Supportive Care (Denosumab)
Number analyzed (Participants) | 21
percent change | -4.28 (7.13)

2. Primary Outcome: Slope in Hip Bone Mineral Density (g/cm^2 Per Day) Regressed on Time in Dual
Description: Parameter estimate of the slope of the regression model of the hip bone mineral density change at day 465 post-HSCT regressed on the enrollment BMD levels.
Time Frame: From the time of enrollment up to 465 days post-HSCT
Population: All treated and eligible patients with measures collected
Measure: Number (95% Confidence Interval); unit: g/cm^2 per day
Arm/Group | Supportive Care (Denosumab)
Number analyzed (Participants) | 21
g/cm^2 per day | 0.04026 [-0.11686 to 0.1973]

3. Primary Outcome: Mean Lumbar Spine Percent Change in Bone Mineral Density (BMD)
Description: Day 0 dual x-ray absorptiometry (DXA) scan and day 465 DXA scan will be compared based on the percent change in BMD in lumbar spine in allogeneic HSCT patients who have experienced either at least 5% BMD loss between baseline (pre- HSCT) and day + 100 post-HSCT, or who have osteopenia or osteoporosis at either the pre-bone marrow transplant or day + 100 DXA scan.
Time Frame: At baseline and 465 days post-HSCT
Population: All treated and eligible patients that had measure taken at day 0 and day 465
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Supportive Care (Denosumab)
Number analyzed (Participants) | 21
percentage change | 0.77 (5.85)

4. Primary Outcome: Mean Total Hip Percent Change in Bone Mineral Density (BMD)
Description: Day 100 dual x-ray absorptiometry (DXA) scan will be compared based on the percent change in BMD in the Total hip in allogeneic HSCT patients who have experienced either at least 5% BMD loss between baseline (pre- HSCT) and day + 100 post-HSCT, or who have osteopenia or osteoporosis at either the pre-bone marrow transplant or day + 100 DXA scan.
Time Frame: At baseline, at time of enrollment (day 100 post-hematopoietic stem cell transplantation [HSCT])
Population: All treated and eligible patients with measure at day 0 and day 100
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Supportive Care (Denosumab)
Number analyzed (Participants) | 29
percentage change | -7.61 (4.54)

5. Primary Outcome: Slope in Lumbar Spine Bone Mineral Density (g/cm^2 Per Day) Regressed on Time in Dual
Description: Parameter estimate of the slope of the regression model of the lumbar spine bone mineral density change at day 465 post-HSCT regressed on the enrollment BMD levels.
Time Frame: From the time of enrollment up to 465 days post-HSCT
Population: All treated and eligible patients with measures collected
Measure: Number (95% Confidence Interval); unit: g/cm^2 per day
Arm/Group | Supportive Care (Denosumab)
Number analyzed (Participants) | 21
g/cm^2 per day | -0.09690 [-0.24883 to 0.05503]

6. Secondary Outcome: Mean Lumbar Spine Percent Change in BMD
Description: Day 100 dual x-ray absorptiometry (DXA) scan will be compared based on the percent change in BMD in the lumbar spine in allogeneic HSCT patients who have experienced either at least 5% BMD loss between baseline (pre- HSCT) and day + 100 post-HSCT, or who have osteopenia or osteoporosis at either the pre-bone marrow transplant or day + 100 DXA scan.
Time Frame: Baseline up to 100 days post-HSCT
Population: All treated and eligible patients with measures at day 0 and day 100
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Supportive Care (Denosumab)
Number analyzed (Participants) | 29
percentage change | -4.04 (5.46)

7. Secondary Outcome: Frequency of Bone Fractures
Description: The number of participants with bone fractures tabulated overall
Time Frame: Up to 1 year post-HSCT
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Denosumab)
Number analyzed (Participants) | 21
Participants | 0

8. Secondary Outcome: Number of Participants That Experienced Any AE
Description: Including but not limited to the following: Injection/hypersensitivity related reactions; osteonecrosis of the jaw; graft versus host disease. Will be assessed according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5 and tabulated by grade.
Time Frame: Up to 30 days
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Supportive Care (Denosumab)
Number analyzed (Participants) | 30
Participants | 7

ADVERSE EVENTS:
Time Frame: AE Time frame - Baseline, weekly until 30 day follow-up.
Arm/Group | Supportive Care (Denosumab)
All-Cause Mortality (participants affected / at risk) | 7/30
Serious Adverse Events (participants affected / at risk) | 5/30
Other Adverse Events (participants affected / at risk) | 2/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Denosumab) (N=30)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Denosumab) (N=30)
Neutrophil count decreased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The targeted sample size was n=114, with n=30 the primary analysis is underpowered. Potential reversal of bone loss might occur over a longer period of time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/32/NCT03925532/Prot_SAP_000.pdf